CLINICAL TRIAL: NCT07382505
Title: Prospective Cohort to Evaluate the Prognostic and Early-Recurrence Detection Performance of Blood-based Minimal Residual Disease (MRD) Testing in Endometrial and Cervical Cancer
Brief Title: Prospective Cohort Study of Minimal Residual Disease(MRD) Testing for Early Recurrence Detection in Endometrial and Cervical Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-Yeol Park, MD, PhD, professor, Asan Medical Center
Other Study IDs: Seoul Asan Medical Center
Record Dates: First submitted 2026-01-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Uterine Neoplasms; Cervical Cancer
Keywords: Endometrial Cancer; Cervical Cancer; Minimal Residual Disease; MRD; Circulating Tumor DNA; Liquid Biopsy
MeSH Terms: conditions — Uterine Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — The study will collect and retain the following biospecimens for the evaluation of Minimal Residual Disease (MRD) and genomic profiling:
  Whole Blood (20 mL): Collected at multiple time points (diagnosis, post-surgery, post-adjuvant therapy, and every 3 months during follow-up).
  Tumor Tissue: Formalin-Fixed Paraffin-Embedded (FFPE) blocks or slides from diagnostic biopsies or surgical specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endometrial cancer cohort: patients diagnosed with endometrial cancer
  Interventions: Genetic: Serial blood collection for MRD testing
- cervical cancer cohort: patients diagnosed with cervical cancer
  Interventions: Genetic: Serial blood collection for MRD testing

INTERVENTIONS:
Genetic: Serial blood collection for MRD testing — Participants will undergo serial peripheral blood collection (approximately 20 mL per visit) at predefined clinical milestones: baseline (diagnosis), post-operative (2-4 weeks after surgery), post-adjuvant therapy (2-4 weeks after completion of chemotherapy or CCRT), and during follow-up surveillance (every 3 months for up to 24 months).
  The collected blood will be used to perform Minimal Residual Disease (MRD) testing by analyzing circulating tumor DNA (ctDNA).
  Archival tumor tissue (FFPE blocks or slides) from initial diagnosis or surgery will also be collected to identify patient-specific somatic mutations for the MRD assay.
  This study is observational and does not involve any changes to the patient's standard of care or medical treatment.

SUMMARY:
This study aims to evaluate the clinical performance of blood-based Minimal Residual Disease (MRD) testing using circulating tumor DNA (ctDNA) in patients with endometrial and cervical cancer. The researchers will investigate whether MRD detection can identify cancer recurrence earlier than current standard imaging or clinical methods (providing a "lead time"). Participants will undergo blood collection at specific time points, including at diagnosis, after surgery, and during regular follow-up visits. The study will also assess the correlation between MRD status and survival outcomes, such as Relapse-Free Survival (RFS) and Overall Survival (OS). The goal is to establish a foundation for personalized treatment strategies based on molecular monitoring.

DETAILED DESCRIPTION:
Despite standard treatments, a significant number of patients with endometrial and cervical cancer experience recurrence. Current monitoring relies on imaging (CT/MRI) and tumor markers (CA-125, SCC-Ag), which often detect recurrence only after a visible tumor mass has formed. This prospective cohort study evaluates the utility of ctDNA-based MRD testing as a high-sensitivity biomarker for early detection.

Study Population and Workflow: A total of 600 participants (300 with endometrial cancer and 300 with cervical cancer) will be enrolled. The study involves the following procedures:

Tumor Tissue Collection: Formalin-fixed paraffin-embedded (FFPE) tissue from surgery or biopsy will be collected for genomic profiling.

Serial Blood Collection: Peripheral blood samples (approximately 20ml) will be collected at:

Baseline (before surgery or CCRT)

Post-operative (within 4 weeks after surgery)

Post-adjuvant therapy (within 4 weeks after completion of chemotherapy or CCRT)

Surveillance (every 3 months for the first 2 years, then every 6 months)

MRD Analysis: Deep sequencing of plasma cell-free DNA (cfDNA) will be performed to track tumor-specific variants.

Objectives: The primary objective is to calculate the "lead time," defined as the interval between the first MRD-positive result and clinical/radiological recurrence. Secondary objectives include evaluating the sensitivity and specificity of the MRD assay and its association with RFS and OS. By comparing MRD dynamics with conventional biomarkers, this study seeks to determine if molecular monitoring can provide a more accurate assessment of a patient's prognosis and risk of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial cancer or cervical cancer.
* Scheduled for or completed standard treatment (Surgery, Adjuvant therapy, or CCRT).
* Provision of written informed consent for study participation and biospecimen collection

Exclusion Criteria:

* Synchronous other malignancies (cancer requiring treatment within the last 5 years).
* Persistent infection or bleeding tendency that makes repeated blood collection unsafe.
* Inability to follow-up or communicate (e.g., due to geographic or cognitive reasons).
* Any condition that the principal investigator deems inappropriate for the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of female patients aged 19 to 79 who have been histologically diagnosed with either endometrial cancer or cervical cancer at Asan Medical Center. This cohort includes patients across various stages of the disease who are scheduled to undergo or have completed standard-of-care treatments, such as radical surgery, adjuvant chemotherapy, radiotherapy, or concurrent chemoradiotherapy (CCRT). The population is designed to represent a real-world clinical setting of gynecologic oncology patients to evaluate the effectiveness of MRD monitoring in predicting recurrence and survival outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of enrollment until the date of first documented recurrence or death from any cause, whichever occurs first, assessed up to 48 months.
  Evaluation of the association between MRD status (detected vs. not detected) and the risk of recurrence or death. MRD will be analyzed as a time-dependent covariate in a Cox proportional hazards model.

SECONDARY OUTCOMES:
Sensitivity and Specificity of MRD Assay | Assessed at specific landmarks (e.g., post-surgery and completion of adjuvant therapy) up to 48 months.
  Evaluation of the diagnostic performance metrics, including sensitivity, specificity, negative predictive value (NPV), and positive predictive value (PPV) of ctDNA-based MRD testing for predicting clinical recurrence.
Overall Survival (OS) | From the date of enrollment until the date of death from any cause, assessed up to 48 months.
  Comparison of the overall survival rate between patients with MRD-positive and MRD-negative results using the Hazard Ratio (HR).

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No